CLINICAL TRIAL: NCT00005151
Title: Pawtucket Heart Health Program
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1022; R01HL023629 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2000-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypercholesterolemia; Hypertension; Obesity; Cerebrovascular Accident; Coronary Disease; Atherosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypercholesterolemia; Hypertension; Obesity; Stroke; Coronary Disease; Atherosclerosis

SUMMARY:
To conduct a community-based research and demonstration project in cardiovascular disease prevention in the town of Pawtucket, Rhode Island. Targeted risk factors included high blood pressure, elevated blood cholesterol, obesity, cigarette smoking, and sedentary living. To evaluate the program, risk factor surveys on a cross-sectional and cohort basis were conducted along with mortality and morbidity surveillance both in Pawtucket and in the non-intervention comparison town of New Bedford, Massachusetts.

DETAILED DESCRIPTION:
BACKGROUND:

The Pawtucket Heart Health Program arose from a concern that the needs of society could not be met through palliative treatment of coronary heart disease. In 1977, a program designed to facilitate rehabilitation and, hopefully, to provide possible secondary preventive measures for patients with symptomatic coronary heart disease was begun. Simultaneously, the conviction grew that the national interest would be served by careful research into whether or not coronary heart disease was preventable through modification of those aspects of individual and group behavior which influenced the major cardiovascular risk factors in free living populations.

The Pawtucket Heart Health Program was designed to foster community ownership and active participation in a culture change process. A population-wide atherosclerosis risk factor reduction was anticipated as a result of applying an independent variable based upon Social Learning Theory. Emphases on individual factors, on physical environmental factors, and on sociocultural influences on behavior were designed to produce persisting risk factor change followed by morbidity - mortality rate reduction for the population of the city.

DESIGN NARRATIVE:

Selection of an intervention community and a control community was carried out early in the design of the Pawtucket Heart Health Program. Census data, as updated through 1975, were used to identify two communities with between 40,000 and 100,000 people and with stability of in-migration and out-migration necessary for long-term follow-up. The two communities were carefully matched for socio-demographic variables.

Both communities underwent baseline random-sample surveys which demonstrated similar levels of cardiovascular risk factors in the populations of each city. Effective community intervention began in 1983. Total intervention was 7.5 years. Specific objectives of the intervention included a six percent reduction in total cholesterol, a 6 mm Hg reduction in systolic blood pressure, a 30 percent relative reduction in active smokers, a two percent reduction in body weight and body mass index, a 2 ml/kg/minute increase in estimated maximal oxygen uptake, and a 15 percent reduction in fatal and non-fatal cardiovascular disease event rates. Educational techniques used by the program included: print, radio and televised messages; small group behavior change programs delivered by trained lay volunteers; community and worksite-based blood pressure reduction, cholesterol and multiple-risk factor screening, counseling and referral events; self-help programs; school curricula; smoking prevention programs; risk behavior change competitions; shelf-labeling in grocery stores and menu-labeling in restaurants to indicate low sodium and low fat foods.

The effectiveness of the program was evaluated by biennial random household risk factor surveys, a morbidity and mortality surveillance system and other methods. In the risk factor survey, households were randomly selected. Within each sampled household, a single respondent was selected from eligible adults. A household interview and testing protocol was administered in the home and includes questions about diet, exercise, smoking, behavior and knowledge of cardiovascular disease. Physiological measures included height, weight, blood pressure, total cholesterol, triglycerides, high-density-lipoprotein bound cholesterol and serum cotinine. A subsample was given a step test to estimate maximum oxygen uptake as a measure of fitness. A second subset completed a Willett diet questionnaire. There were five cross-sectional household surveys of approximately 2,800 individuals per survey. The initial cross-sectional survey was converted to a cohort survey for measurement again in 1986-1987 and in 1988-1989. The third cross-sectional survey was also converted to a cohort survey for simultaneous measurement with the 1987-1988 and 1989-1990 cross-sectional samples.

Both communities were screened for morbidity and case-fatality rates for coronary heart disease and stroke. Morbidity and mortality data were obtained from seven area hospitals and the State Health Departments of Rhode Island and Massachusetts. Outcome criteria were developed collaboratively by the Pawtucket Heart Health Program, the Stanford Five-City Multifactor Risk Reduction Study, and the Minnesota Heart Health Program, to maximize the scientific value of the conclusions drawn from the three studies and to allow pooling of final data. Surveillance was complete for 1980 to 1983 and continued through 1993.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1980-08; Study Completion 1997-07 (Actual)

REFERENCES:
- [Background] Gans KM, Lapane KL, Lasater TM, Carleton RA. Effects of intervention on compliance to referral and lifestyle recommendations given at cholesterol screening programs. Am J Prev Med. 1994 Sep-Oct;10(5):275-82. PMID 7848670
- [Background] Crowley JP, Metzger J, Assaf A, Carleton RC, Merrill E, Valeri CR. Low density lipoprotein cholesterol and whole blood viscosity. Ann Clin Lab Sci. 1994 Nov-Dec;24(6):533-41. PMID 7847781
- [Background] Derby CA, Hume AL, McPhillips JB, Barbour MM, Carleton RA. Prior and current health characteristics of postmenopausal estrogen replacement therapy users compared with nonusers. Am J Obstet Gynecol. 1995 Aug;173(2):544-50. doi: 10.1016/0002-9378(95)90280-5. PMID 7645633
- [Background] Carleton RA, Lasater TM, Assaf AR, Feldman HA, McKinlay S. The Pawtucket Heart Health Program: community changes in cardiovascular risk factors and projected disease risk. Am J Public Health. 1995 Jun;85(6):777-85. doi: 10.2105/ajph.85.6.777. PMID 7762709
- [Background] Carleton RA, Lasater TM, Assaf AR. The Pawtucket Heart Health Program: progress in promoting health. R I Med. 1995 Mar;78(3):74-7. No abstract available. PMID 7734757
- [Background] Derby CA, Lasater TM, Vass K, Gonzalez S, Carleton RA. Characteristics of smokers who attempt to quit and of those who recently succeeded. Am J Prev Med. 1994 Nov-Dec;10(6):327-34. PMID 7880551
- [Background] Coronary-prone behavior and coronary heart disease: a critical review. The review panel on coronary-prone behavior and coronary heart disease. Circulation. 1981 Jun;63(6):1199-215. doi: 10.1161/01.cir.63.6.1199. PMID 7014026
- [Background] Thompson PD, Funk EJ, Carleton RA, Sturner WQ. Incidence of death during jogging in Rhode Island from 1975 through 1980. JAMA. 1982 May 14;247(18):2535-8. PMID 6978411
- [Background] Siconolfi SF, Cullinane EM, Carleton RA, Thompson PD. Assessing VO2max in epidemiologic studies: modification of the Astrand-Rhyming test. Med Sci Sports Exerc. 1982;14(5):335-8. PMID 7154887
- [Background] Carleton RA. Criterion for cholesterol norms--healthy or statistical? Am J Clin Pathol. 1983 Mar;79(3):402. doi: 10.1093/ajcp/79.3.402. No abstract available. PMID 6829508
- [Background] Carleton RA, Lasater TM. Coronary heart disease and human behavior. Prev Med. 1983 Sep;12(5):610-8. doi: 10.1016/0091-7435(83)90217-7. PMID 6657626
- [Background] Siconolfi SF, Carleton RA, Elder JP, Bouchard PA: Hypotension After Exercise and Relaxation. In: Canto RC (Ed), Clinical Sports Medicine, Collamore Press, Lexington, Mass, Chapter 11, 1983
- [Background] Hume AL, Barbour MM, Willey CJ, Assaf AR, Lapane KL, Carleton RA. Changing trends in antihypertensive therapy in two New England communities during the 1980s. Pharmacotherapy. 1993 May-Jun;13(3):244-51. PMID 8100629
- [Background] McPhillips JB, Eaton CB, Gans KM, Derby CA, Lasater TM, McKenney JL, Carleton RA. Dietary differences in smokers and nonsmokers from two southeastern New England communities. J Am Diet Assoc. 1994 Mar;94(3):287-92. doi: 10.1016/0002-8223(94)90370-0. PMID 8120293
- [Background] Reynes JF, Lasater TM, Feldman H, Assaf AR, Carleton RA. Education and risk factors for coronary heart disease: results from a New England community. Am J Prev Med. 1993 Nov-Dec;9(6):365-71. PMID 8311986
- [Background] Assaf AR, Lapane KL, McKenney JL, Carleton RA. Possible influence of the prospective payment system on the assignment of discharge diagnoses for coronary heart disease. N Engl J Med. 1993 Sep 23;329(13):931-5. doi: 10.1056/NEJM199309233291307. PMID 8361508
- [Background] Barbour MM, Hume AL, Assaf AR, Carleton RA. The drug data base of the Pawtucket Heart Health Program: development and description. Pharmacotherapy. 1993 May-Jun;13(3):239-43. PMID 8321737
- [Background] Derby CA, Hume AL, Barbour MM, McPhillips JB, Lasater TM, Carleton RA. Correlates of postmenopausal estrogen use and trends through the 1980s in two southeastern New England communities. Am J Epidemiol. 1993 May 15;137(10):1125-35. doi: 10.1093/oxfordjournals.aje.a116616. PMID 8317442
- [Background] Hume AL, Barbour MM, Lapane KL, Assaf AR, Carleton RA. Prevalence and descriptors of aspirin use as an antiplatelet agent in two New England communities. Ann Pharmacother. 1993 Apr;27(4):442-4. doi: 10.1177/106002809302700409. PMID 8477120
- [Background] Gans KM, Jack B, Lasater TM, Lefebvre RC, McQuade W, Carleton RA. Changing physicians' attitudes, knowledge, and self-efficacy regarding cholesterol screening and management. Am J Prev Med. 1993 Mar-Apr;9(2):101-6. PMID 8471266
- [Background] McKinlay SM, Kipp DM, Johnson P, Downey K, Carleton RA: A Field Approach for Obtaining Physiological Measures in Surveys of General Populations: Response Rates, Reliability, and Costs. Health Survey Research Methods: Proceedings of the Fourth Conference on Health Survey Research Methods. Washington, DC, 1982. DHHS Pub. No. (PHS) 84-3346, 1984
- [Background] Siconolfi SF, Garber CE, Baptist GD, Cooper FS, Carleton RA. Circulatory effects of mental stress during exercise in coronary artery disease patients. Clin Cardiol. 1984 Aug;7(8):441-4. doi: 10.1002/clc.4960070804. PMID 6467695
- [Background] Siconolfi SF, Carleton RA, Lasater TM: Relationship Between Physical Activity Questionnaire and Maximal Oxygen Uptake. Circulation, Supplement, October, 1984
- [Background] Sennett LL, Peterson G, Elder JP, Lasater TM, Carleton RA: A Community-Based Approach to Weight Loss: The Pawtucket 'Weigh-In.' Chapter in Clinical Sports Medicine, Third Edition, Canto RC (Ed), Collamore Press, Lexington, Mass, in Press, 1985
- [Background] Elder JP, Artz LM, Beaudin P, Carleton RA, Lasater TM, Peterson G, Rodrigues A, Guadagnoli E, Velicer WF. Multivariate evaluation of health attitudes and behaviors: development and validation of a method for health promotion research. Prev Med. 1985 Jan;14(1):34-54. doi: 10.1016/0091-7435(85)90019-2. PMID 4034513
- [Background] Siconolfi SF, Lasater TM, McKinlay S, Boggia P, Carleton RA. Physical fitness and blood pressure: the role of age. Am J Epidemiol. 1985 Sep;122(3):452-7. doi: 10.1093/oxfordjournals.aje.a114126. PMID 4025294
- [Background] Siconolfi SF, Lasater TM, Snow RC, Carleton RA. Self-reported physical activity compared with maximal oxygen uptake. Am J Epidemiol. 1985 Jul;122(1):101-5. doi: 10.1093/oxfordjournals.aje.a114068. PMID 4014188
- [Background] Siconolfi SF, Garber CE, Lasater TM, Carleton RA. A simple, valid step test for estimating maximal oxygen uptake in epidemiologic studies. Am J Epidemiol. 1985 Mar;121(3):382-90. doi: 10.1093/oxfordjournals.aje.a114010. PMID 4014128
- [Background] Elder JP, McGraw SA, Lasater TM, Peterson G, Ferreira A, Carleton RA, Longpre H, Harden E: Gemeindeweite Praevention von Herzkrankheitten in den U.S.A.: der Pawtucket-Experiment. Pravention (FRG), 1986
- [Background] Elder JP, McKenna CA, Lazieh M, Ferreira A, Lasater TM, Carleton RA. The use of volunteers in mass screening for high blood pressure. Am J Prev Med. 1986 Sep-Oct;2(5):268-72. PMID 3453190
- [Background] Schwertfeger R, Elder JP, Cooper R, Lasater TM, Carleton R. The use of telemarketing in the community-wide prevention of heart disease: the Pawtucket Heart Health Program. J Community Health. 1986 Fall;11(3):172-80. doi: 10.1007/BF01338798. PMID 3793968
- [Background] Siconolfi SF, Lasater TM, Elder JP, Garber CE, Carleton RA: Normal Blood Pressure Reactivity to Mental Stress in Borderline Hypertensive Patients. J Cardiac Rehab, 6:383-398, 1986
- [Background] Lefebvre RC, Peterson GS, McGraw SA, Lasater TM, Sennett L, Kendall L, Carleton RA. Community intervention to lower blood cholesterol: the "Know Your Cholesterol" campaign in Pawtucket, Rhode Island. Health Educ Q. 1986 Summer;13(2):117-29. doi: 10.1177/109019818601300202. PMID 3721878
- [Background] Elder JP, McGraw SA, Abrams DB, Ferreira A, Lasater TM, Longpre H, Peterson GS, Schwertfeger R, Carleton RA. Organizational and community approaches to community-wide prevention of heart disease: the first two years of the Pawtucket Heart Health Program. Prev Med. 1986 Mar;15(2):107-17. doi: 10.1016/0091-7435(86)90081-2. PMID 3714665
- [Background] Peterson G, Elder JP, Knisley PM, Colby JC, Beaudin P, DeBlois D, Carleton RA. Developing strategies for food vendor intervention: the first step. J Am Diet Assoc. 1986 May;86(5):659-61. No abstract available. PMID 3700928
- [Background] Peterson GS, Lefebvre RC, Ferreira A, Sennett L, Lazieh M, Carleton RA: Strategies for Cholesterol Lowering at the Worksite, J Nutr Educ, 18(1), 1986
- [Background] McKinlay SM, McGraw SA, Assaf AR, Kipp DM, Carleton RA: An Innovative Approach to the Evaluation of Large Community Programs. In: Baum A, Herd JA, (Eds). Perspectives in Behavioral Medicine, Volume 3. Academic Press, Inc. New York, 1987
- [Background] Carleton RA, Lasater TM. Primary prevention of coronary heart disease: a challenge for behavioral medicine. Circulation. 1987 Jul;76(1 Pt 2):I124-9. PMID 3297395
- [Background] Elder JP, Abrams DB, Beaudin P, Carleton RA, Lasater TM, Lazieh M, Peterson G, Schwertfeger R: Behavioral Community Psychology and the Prevention of Heart Disease: Community Level Applications of the Pawtucket Heart Health Program. In: Baum A, Herd A, (Eds). Perspectives in Behavioral Medicine, Volume 3. Academic Press, Inc. New York, 1987
- [Background] Lasater TM, Elder JP, Carleton RA, Abrams DB. The Pawtucket Heart Health Program: Prospects and Process. In: Baum A, Herd JA (Eds). Perspectives in Behavioral Medicine, Volume 3. Academic Press, Inc. New York, 1987
- [Background] Harden EA, Lefebvre RC, Fuchs V, Lasater TM, Carleton RA: Telemarketing for Health Promotion. Am J Prev Med, 1987
- [Background] Lefebvre RC, Lasater TM, Carleton RA, Peterson G. Theory and delivery of health programming in the community: the Pawtucket Heart Health Program. Prev Med. 1987 Jan;16(1):80-95. doi: 10.1016/0091-7435(87)90008-9. PMID 3823012
- [Background] Nelson DJ, et al: A Campaign Strategy for Weight Loss at Worksites. Health Educ Res: Theory and Practice, 2:27-31, 1987
- [Background] Lefebvre RC. Primary prevention of coronary heart disease: a review of multifactor prevention trials. Prog Behav Modif. 1987;21:45-85. No abstract available. PMID 3108868
- [Background] Lasater TM, Lefebvre RC, Assaf AR, Saritelli AL, Carleton RA. Rapid measurement of blood cholesterol: evaluation of a new instrument. Am J Prev Med. 1987 Nov-Dec;3(6):311-6. PMID 3452369
- [Background] Lefebvre RC, Harden EA, Rakowski W, Lasater TM, Carleton RA. Characteristics of participants in community health promotion programs: four-year results. Am J Public Health. 1987 Oct;77(10):1342-4. doi: 10.2105/ajph.77.10.1342. PMID 3631372
- [Background] Elder JP, McGraw SA, Rodrigues A, Lasater TM, Ferreira A, Kendall L, Peterson G, Carleton RA. Evaluation of two community-wide smoking cessation contests. Prev Med. 1987 Mar;16(2):221-34. doi: 10.1016/0091-7435(87)90086-7. PMID 3588563
- [Background] Assaf AR, Banspach SW, Lasater TM, McKinlay SM, Carleton RA. The Pawtucket Heart Health Program: II. Evaluation strategies. R I Med J (1976). 1987 Dec;70(12):541-6. No abstract available. PMID 3480550
- [Background] Carleton RA, Lasater TM, Assaf A, Lefebvre RC, McKinlay SM. The Pawtucket Heart Health Program: I. An experiment in population-based disease prevention. R I Med J (1976). 1987 Dec;70(12):533-8. No abstract available. PMID 3480549
- [Background] Colby JJ, Elder JP, Peterson G, Knisley PM, Carleton RA. Promoting the selection of healthy food through menu item description in a family-style restaurant. Am J Prev Med. 1987 May-Jun;3(3):171-7. PMID 3452355
- [Background] Lefebvre RC, Lasater TM, Assaf AR, Carleton RA. Pawtucket Heart Health Program: the process of stimulating community change. Scand J Prim Health Care Suppl. 1988;1:31-7. PMID 3227200
- [Background] Block L, Banspach SW, Gans K, Harris C, Lasater TM, Lefebvre RC, Carleton RA. Impact of public education and continuing medical education on physician attitudes and behavior concerning cholesterol. Am J Prev Med. 1988 Sep-Oct;4(5):255-60. PMID 3224002
- [Background] Lefebvre RC, Harden EA, Zompa B. The Pawtucket Heart Health Program. III. Social marketing to promote community health. R I Med J (1976). 1988 Jan;71(1):27-30. No abstract available. PMID 3422499
- [Background] Lasater TM, Lefebvre RC, Carleton RA. The Pawtucket Heart Health Program. IV. Community level programming for heart health. R I Med J (1976). 1988 Jan;71(1):31-4. No abstract available. PMID 3422500
- [Background] Lasater TM, Carleton RA, Lefebvre RC. The Pawtucket Heart Health Program. V. Utilizing community resources for primary prevention. R I Med J (1976). 1988 Feb;71(2):63-7. No abstract available. PMID 3162330
- [Background] Lefebvre RC, Hursey KG, Carleton RA. Labeling of participants in high blood pressure screening programs. Implications for blood cholesterol screenings. Arch Intern Med. 1988 Sep;148(9):1993-7. PMID 3046540
- [Background] Lefebvre RC, Lasater TH, McKinlay SM, Gans KM, Walker N, Carleton RA. Performance characteristics of a blood cholesterol measuring instrument used in screening programs. Public Health Rep. 1989 May-Jun;104(3):266-70. PMID 2498976
- [Background] McKinlay SM, Carleton RA, McKenney JL, Assaf AR. A new approach to surveillance for acute myocardial infarction: reproducibility and cost efficiency. Int J Epidemiol. 1989 Mar;18(1):67-75. doi: 10.1093/ije/18.1.67. PMID 2498218
- [Background] Niknian M, McKinlay SM, Rakowski W, Carleton RA. A comparison of perceived and objective CVD risk in a general population. Am J Public Health. 1989 Dec;79(12):1653-4. doi: 10.2105/ajph.79.12.1653. PMID 2817194
- [Background] Gans KM, Levin S, Lasater TM, Sennett LL, Maroni A, Ronan A, Carleton RA. Heart healthy cook-offs in home economics classes: an evaluation with junior high school students. J Sch Health. 1990 Mar;60(3):99-102. doi: 10.1111/j.1746-1561.1990.tb05409.x. PMID 2319756
- [Background] Lefebvre RC, Gubata P, Ronan A, Carleton RA. Variation in the Reflotron method of cholesterol measurement. Am J Cardiol. 1990 Apr 1;65(13):916-7. doi: 10.1016/0002-9149(90)91437-b. No abstract available. PMID 2321542
- [Background] Hunt MK, Lefebvre RC, Hixson ML, Banspach SW, Assaf AR, Carleton RA. Pawtucket Heart Health Program point-of-purchase nutrition education program in supermarkets. Am J Public Health. 1990 Jun;80(6):730-2. doi: 10.2105/ajph.80.6.730. PMID 2343964
- [Background] Linnan LA, Harden EA, Bucknam L, Carleton RA. Marketing cardiovascular disease risk reduction programs at the workplace. The Pawtucket Heart Health Program experience. AAOHN J. 1990 Sep;38(9):409-18. PMID 2397012
- [Background] Rakowski W, Lefebvre RC, Assaf AR, Lasater TM, Carleton RA. Health practice correlates in three adult age groups: results from two community surveys. Public Health Rep. 1990 Sep-Oct;105(5):481-91. PMID 2120725
- [Background] Lefebvre RC, Cobb GD, Goreczny AJ, Carleton RA. Efficacy of an incentive-based community smoking cessation program. Addict Behav. 1990;15(5):403-11. doi: 10.1016/0306-4603(90)90026-t. PMID 2248113
- [Background] Linnan LA, Gans KM, Hixson ML, Mendes E, Longpre H, Carleton RA. Training health professionals and lay volunteers to deliver cholesterol screening and education programs. Public Health Rep. 1990 Nov-Dec;105(6):589-98. PMID 2124360
- [Background] Rakowski W, Assaf AR, Lefebvre RC, Lasater TM, Niknian M, Carleton RA. Information-seeking about health in a community sample of adults: correlates and associations with other health-related practices. Health Educ Q. 1990 Winter;17(4):379-93. doi: 10.1177/109019819001700403. PMID 2262319
- [Background] Assaf AR, Banspach SW, Lasater TM, Ramsey J, Tidwell RJ, Carleton RA. The FPbase microcomputer system for managing community health screening and intervention data bases. Public Health Rep. 1992 Nov-Dec;107(6):695-700. PMID 1333621
- [Background] DelPrete LR, Caldwell M, English C, Banspach SW, Lefebvre C. Self-reported and measured weights and heights of participants in community-based weight loss programs. J Am Diet Assoc. 1992 Dec;92(12):1483-6. PMID 1452961
- [Background] Jack BW, Gans KM, McQuade W, Culpepper L, Lasswell A, Hume AL, Dowling PT, Carleton RA. A successful physician training program in cholesterol screening and management. Prev Med. 1991 May;20(3):364-77. doi: 10.1016/0091-7435(91)90035-3. PMID 1862058
- [Background] Lasater TM, Sennett LL, Lefebvre RC, DeHart KL, Peterson G, Carleton RA. Community-based approach to weight loss: the Pawtucket "weigh-in". Addict Behav. 1991;16(3-4):175-81. doi: 10.1016/0306-4603(91)90010-f. PMID 2063705
- [Background] Carleton RA, Sennett L, Gans KM, Levin S, Lefebvre C, Lasater TM. The Pawtucket Heart Health Program. Influencing adolescent eating patterns. Ann N Y Acad Sci. 1991;623:322-6. doi: 10.1111/j.1749-6632.1991.tb43741.x. PMID 2042840
- [Background] Niknian M, Linnan LA, Lasater TM, Carleton RA. Use of population-based data to assess risk factor profiles of blue and white collar workers. J Occup Med. 1991 Jan;33(1):29-36. doi: 10.1097/00043764-199101000-00010. PMID 1995799
- [Background] Niknian M, Lefebvre RC, Carleton RA. Are people more health conscious? A longitudinal study of one community. Am J Public Health. 1991 Feb;81(2):205-7. doi: 10.2105/ajph.81.2.205. PMID 1990861
- [Background] Eaton CB, Lapane KL, Garber CA, Assaf AR, Lasater TM, Carleton RA. Sedentary lifestyle and risk of coronary heart disease in women. Med Sci Sports Exerc. 1995 Nov;27(11):1535-9. PMID 8587490
- [Background] McKenney JL, Lapane KL, Assaf AR, Carleton RA. The association between perceived risk and actual cardiovascular disease. Epidemiology. 1995 Nov;6(6):612-6. doi: 10.1097/00001648-199511000-00009. PMID 8589093
- [Background] Assaf AR, Helmert U, Lasater TL, Carleton RA, Greiser E. Measuring cardiovascular disease risk factor levels: international comparisons between Bremen-north/west (Germany) and two southeastern New England (USA) cities. Soz Praventivmed. 1995;40(4):218-29. doi: 10.1007/BF01354476. PMID 8525711
- [Background] Eaton CB, McPhillips JB, Gans KM, Garber CE, Assaf AR, Lasater TM, Carleton RA. Cross-sectional relationship between diet and physical activity in two southeastern New England communities. Am J Prev Med. 1995 Jul-Aug;11(4):238-44. PMID 7495600
- [Background] Lapane KL, Zierler S, Lasater TM, Barbour MM, Carleton R, Hume AL. Is the use of psychotropic drugs associated with increased risk of ischemic heart disease? Epidemiology. 1995 Jul;6(4):376-81. doi: 10.1097/00001648-199507000-00008. PMID 7548344
- [Background] Derby CA, Feldman HA, Bausserman LL, Parker DR, Gans KM, Carleton RA. HDL cholesterol: trends in two southeastern New England communities, 1981-1993. Ann Epidemiol. 1998 Feb;8(2):84-91. doi: 10.1016/s1047-2797(97)00130-0. PMID 9491932
- [Background] Winkleby MA, Feldman HA, Murray DM. Joint analysis of three U.S. community intervention trials for reduction of cardiovascular disease risk. J Clin Epidemiol. 1997 Jun;50(6):645-58. doi: 10.1016/s0895-4356(97)00020-6. PMID 9250263
- [Background] Parker DR, Gonzalez S, Derby CA, Gans KM, Lasater TM, Carleton RA. Dietary factors in relation to weight change among men and women from two southeastern New England communities. Int J Obes Relat Metab Disord. 1997 Feb;21(2):103-9. doi: 10.1038/sj.ijo.0800373. PMID 9043963
- [Background] Derby CA, Lapane KL, Hume AL, Babour MM, Carleton RA. Is cigarette smoking an effect modifier of the relation between antihypertensive therapy and blood lipids? Epidemiology. 1997 Jan;8(1):48-54. doi: 10.1097/00001648-199701000-00008. PMID 9116095
- [Background] Hume AL, Barbour MM, Lapane KL, Flint PM, Carleton RA. Correlates of oral contraceptive use in two New England communities: 1981-1993. Pharmacotherapy. 1996 Nov-Dec;16(6):1173-8. PMID 8947992
- [Background] Parker DR, Derby CA, Usner DW, Gonzalez S, Lapane KL, Carleton RA. Self-reported alcohol intake using two different question formats in southeastern New England. Int J Epidemiol. 1996 Aug;25(4):770-4. doi: 10.1093/ije/25.4.770. PMID 8921455
- [Background] Parker DR, McPhillips JB, Lapane KL, Lasater TM, Carleton RA. Nutrition and health practices of diabetic and nondiabetic men and women from two southeastern New England communities. Nutr Health. 1995;10(3):255-68. doi: 10.1177/026010609501000309. PMID 8684734
- [Background] Parker DR, McPhillips JB, Derby CA, Gans KM, Lasater TM, Carleton RA. High-density-lipoprotein cholesterol and types of alcoholic beverages consumed among men and women. Am J Public Health. 1996 Jul;86(7):1022-7. doi: 10.2105/ajph.86.7.1022. PMID 8669505
- [Background] Flint PM, Lapane KL, Barbour MM, Derby CA, Carleton RA, Hume AL. Cardiovascular risk profiles of oral contraceptive users and nonusers: a population-based study. Prev Med. 1995 Nov;24(6):586-90. doi: 10.1006/pmed.1995.1093. PMID 8610082
- [Background] Lapane KL, Zierler S, Lasater TM, Stein M, Barbour MM, Hume AL. Is a history of depressive symptoms associated with an increased risk of infertility in women? Psychosom Med. 1995 Nov-Dec;57(6):509-13; discussion 514-6. doi: 10.1097/00006842-199511000-00001. PMID 8600476
- [Background] Assaf AR, Lapane KL, McKenney JL, McKinlay S, Carleton RA. Coronary heart disease surveillance: field application of an epidemiologic algorithm. J Clin Epidemiol. 2000 Apr;53(4):419-26. doi: 10.1016/s0895-4356(99)00183-3. PMID 10785573
- [Background] Derby CA, Lapane KL, Feldman HA, Carleton RA. Trends in validated cases of fatal and nonfatal stroke, stroke classification, and risk factors in southeastern New England, 1980 to 1991 : data from the Pawtucket Heart Health Program. Stroke. 2000 Apr;31(4):875-81. doi: 10.1161/01.str.31.4.875. PMID 10753991
- [Background] Derby CA, Lapane KL, Feldman HA, Carleton RA. Sex-specific trends in validated coronary heart disease rates in southeastern New England, 1980-1991. Am J Epidemiol. 2000 Feb 15;151(4):417-29. doi: 10.1093/oxfordjournals.aje.a010222. PMID 10695601
- [Background] Eaton CB, Lapane KL, Garber CE, Gans KM, Lasater TM, Carleton RA. Effects of a community-based intervention on physical activity: the Pawtucket Heart Health Program. Am J Public Health. 1999 Nov;89(11):1741-4. doi: 10.2105/ajph.89.11.1741. PMID 10553400
- [Background] Gans KM, Assmann SF, Sallar A, Lasater TM. Knowledge of cardiovascular disease prevention: an analysis from two New England communities. Prev Med. 1999 Oct;29(4):229-37. doi: 10.1006/pmed.1999.0532. PMID 10547047
- [Background] Parker DR, Lapane KL, Lasater TM, Carleton RA. Short stature and cardiovascular disease among men and women from two southeastern New England communities. Int J Epidemiol. 1998 Dec;27(6):970-5. doi: 10.1093/ije/27.6.970. PMID 10024190